CLINICAL TRIAL: NCT06731218
Title: A Single-Center, Single-Arm, Open-Label Phase I Clinical Trial Evaluating the Safety and Efficacy of RGB-5088 Islet Cell Injection in the Treatment of Type 1 Diabetes Mellitus
Brief Title: Phase I Clinical Study to Evaluate the Safety and Efficacy of RGB-5088 in Patients With Type 1 Diabetes Mellitus
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Hangzhou Reprogenix Bioscience, Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RGB-5088-01
Record Dates: First submitted 2024-12-09; First posted 2024-12-12 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Diabetes Mellitus, Type 1; Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- RGB-5088 (Experimental): Transplantation under the anterior rectus sheath
  Interventions: Biological: RGB-5088

INTERVENTIONS:
Biological: RGB-5088 — Transplantation under the anterior rectus sheath

SUMMARY:
This Phase I clinical trial is a single-center, single-arm, open-label study aimed at evaluating the safety and therapeutic efficacy of RGB-5088 islet cell transplantation in patients with Type 1 Diabetes Mellitus.

ELIGIBILITY:
Key Inclusion Criteria:

* Age: 18-60 years old (including 18 and 60 years old), male and female;
* Type 1 diabetes patients (including those who have received organ transplantation such as liver and kidney);
* Stimulated C-peptide < 0.3 ng/mL;
* The patient had at least one severe hypoglycemia within 12 months before being included in the project

Key Exclusion Criteria:

* Type 2 diabetes patients;
* Untreated proliferative diabetes retinopathy;
* Serious heart disease;
* Serious gastrointestinal dysfunction ；
* Serious psychological diseases；
* Any history of malignancy;
* Have a history of tobacco, alcohol and drug abuse;
* For female subjects: pregnancy test positive, lactation or unwilling to use effective contraceptive measures during the study period, male patients: intent to procreate or unwilling to use effective contraceptive measures during the study period.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-02-17 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2031-12-31 (Estimated)

PRIMARY OUTCOMES:
Safety as assessed by number of subjects with adverse events | From RGB-5088 transplantation to one year later
Proportion of subjects with HbA1c ≤ 6.5% and free of severe hypoglycemic events | From 90 days to 365 days after RGB-5088 transplantation

SECONDARY OUTCOMES:
Safety as assessed by number of subjects with adverse events | From RGB-5088 transplantation to end of study (up to 5 years)
Proportion of subjects who are insulin independent | From 90 days to end of study (up to 5 years)
Proportion of subjects with HbA1c ≤ 6.5% and free of severe hypoglycemic events | From 90 days to end of study (up to 5 years)

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin First Center Hospital, Tianjin, Tianjin Municipality, China